CLINICAL TRIAL: NCT02103946
Title: Serratus Anterior Muscle Plane Block Versus Paravertebral Block for Breast Cancer Resections.
Brief Title: Serratus Anterior Plane Block Versus Paravertebral Block for Postmastectomy Analgesia
Acronym: SAM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ghada M N Bashandy, Dr, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI- Cairo
Record Dates: First submitted 2014-03-04; First posted 2014-04-04 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer; Acute Pain
Keywords: serratus; paravertebral; breast; cancer; axilla
MeSH Terms: conditions — Breast Neoplasms; Acute Pain; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Serratus anterior muscle plane block (Active Comparator): Serratus anterior muscle plane block with general anesthesia MARCAINE® 0.25%w/v solution for injection. DIPRIVAN® (propofol), 2 to 2.5 mg/kg NIMBEX® (cisatracurium besylate) Injection, 0.15-0.2 mg\Kg Fentanyl, 1-2 mic\Kg Paracetamol, 1000 mg\6 hours Fam® (Ketorolac), 30 mg
  Interventions: Procedure: Serratus Anterior Muscle Plane block (SAM block)
- Paravertebral block (Active Comparator): Paravertebral block with general anesthesia. MARCAINE® 0.25%w/v solution for injection. DIPRIVAN® (propofol), 2 to 2.5 mg/kg NIMBEX® (cisatracurium besylate) Injection, 0.15-0.2 mg\Kg Fentanyl, 1-2 mic\Kg Paracetamol, 1000 mg\6 hours Fam® (Ketorolac), 30 mg
  Interventions: Procedure: Paravertebral Block

INTERVENTIONS:
Procedure: Serratus Anterior Muscle Plane block (SAM block) — The US probe is placed in the mid-axillary line at level of the 6th intercostal space. From caudal to cranial, an in-plane approach, the block needle is inserted until the tip is placed between SAM and intercostal muscles and the LA injection will be visualized in real-time. The injection usually consists of 0.4ml/kg of bupivacaine 0.25% plus adrenaline (5ug/ml). Intraoperatively, all subjects will receive a general anesthetic using inhaled anesthetic and oxygen. Intravenous fentanyl will be administered for cardiovascular stability to noxious stimuli.For postoperative analgesia, all subjects will receive oral acetaminophen. Patients will receive a ketorolac IV injection then morphine as a rescue analgesic for breakthrough pain.
  Other Names: Serratus anterior block; intercostal nerve block
  Arms: Serratus anterior muscle plane block
Procedure: Paravertebral Block — After skin preparation and sterile draping applied. Target paravertebral space will be located using US guidance. The paravertebral space between the third and fourth thoracic vertebrae will be identified in a parasagittal view approximately 3 cm lateral to midline on the side of surgery. A local anesthetic skin wheal will be raised caudal to the ultrasound transducer. A 17-gauge, Tuohy-tip needle will be inserted through the skin wheal in-plane beneath the ultrasound transducer and directed to the paravertebral space. Normal saline (5 mL) will be injected via the needle to help identify the paravertebral space and observe the pleura being displaced anteriorly. 0.4 ml\kg of 0.25% Bupivacaine with epinephrine, 5 μg/mL, will be slowly injected with gentle aspiration every 3 mL.
  Other Names: Thoracic Paravertebral block
  Arms: Paravertebral block

SUMMARY:
ًًًُُُُThe investigators are testing the efficacy of a new novel technique; serratus anterior plane block, for preventing postoperative pain after breast surgery for cancer. This block will be compared with the well-established paravertebral block.

DETAILED DESCRIPTION:
Paravertebral block (PVB) can be considered as a well-established option to provide anesthesia and postoperative analgesia during breast surgery. For patients receiving a PVB alone or in combination with general anesthesia significant lower resting, evoked and worst pain scores compared with other analgesic treatment strategies indicating that a PVB provides improved postoperative pain control in patients undergoing breast surgery. Furthermore, there might be a reduced need for postoperative opioid requirements and consecutively a decrease in opioid-induced adverse effects in patients receiving a PVB. Anyways there are always fear of pleural injury and pneumothorax in addition to epidural and intrathecal spread of the block. A novel newly introduced field block has been described recently to block the hemithorax under ultrasound guidance that is the Serratus Anterior Muscle Plane SAM block. Still this technique to the investigators knowledge is not tried in randomized clinical studies. The aim of this study is to find out that this new technique is comparable to PVB in patients undergoing breast surgeries with or without axillary node dissection.

ELIGIBILITY:
Inclusion Criteria:

* unilateral mastectomy with or without axillary lymph node dissection.
* American Society of Anesthesia (ASA) I&II

Exclusion Criteria:

* morbid obesity (body mass index > 40 kg/m2);
* renal insufficiency (creatinine > 1.5 mg/dL),
* current chronic analgesic therapy (daily use > 4 weeks),
* a history of opioid dependence, pregnancy,
* inability to communicate with the investigators or hospital staff,
* American Society of Anesthesia (ASA) III-IV

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
pain relief | first postoperative day
  reduction of pain intensities in the first postoperative day after breast surgery for cancer.

SECONDARY OUTCOMES:
opioid consumption | intraoperative and first postoperative day
  intraoperative and postoperative opioid consumption

OTHER OUTCOMES:
patient satisfaction | first week after surgery
  measure patient satisfaction a week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ghada MN Bashandy, MD, Principal Investigator — Lecturer of anesthesia & pain relief
Locations (1):
- National Cancer Institute, Cairo, Kasr Alainy, Egypt

REFERENCES:
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Mendoza TR, Chen C, Brugger A, Hubbard R, Snabes M, Palmer SN, Zhang Q, Cleeland CS. The utility and validity of the modified brief pain inventory in a multiple-dose postoperative analgesic trial. Clin J Pain. 2004 Sep-Oct;20(5):357-62. doi: 10.1097/00002508-200409000-00011. PMID 15322443
- [Result] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- See also: Serratus plane block: a novel ultrasound-guided thoracic wall nerve block — http://onlinelibrary.wiley.com/doi/10.1111/anae.12344/pdf